CLINICAL TRIAL: NCT05539781
Title: Change of Hemodynamics and Cerebral Functions After Carotid Artery Revascularization
Acronym: HALO
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HALO
Record Dates: First submitted 2022-08-30; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-05

CONDITIONS: Carotid Artery Diseases; Carotid Artery Stenosis; Cerebrovascular; Disorder, Arteriosclerotic; Cardiovascular Diseases; Nervous System Diseases
Keywords: carotid endarterectomy; carotid stenting; computational fluid dynamic; cognitive function; medical therapy
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Intracranial Arteriosclerosis; Cardiovascular Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The majority (>80%) of strokes are of ischemic etiology, of which ≈15% to 20% are attributable to atherosclerosis of the extracranial carotid arteries. The primary goal in carotid artery revascularization is to prevent stroke in patients with carotid artery stenosis. Treatment options including carotid endarterectomy (CEA) and carotid artery stenting (CAS). Hence, the investigators aim to compare carotid artery stenting (CAS) with carotid endarterectomy (CEA) in terms of long-term prognostic endpoints. Also, CEA and CAS result in different postoperative geometric features of carotid arteries that entail relevant modifications of rheological parameters, that may be associated with the risk of local complications and carotid artery restenosis. Finally, long-term and sustained cognitive benefits after carotid artery revascularization need further research and evidence.

DETAILED DESCRIPTION:
Hypothesis and Significance: We hypothesize that hemodynamically changes after carotid artery revascularization influence the cerebral function or carotid artery patency. If cognitive improvement or impairment and carotid artery restenosis can be demonstrated relate to hemodynamic remodeling in these patients, then we will have established a new prognostic factor for carotid revascularization independent of the existing study.

Specific Aim: 1) To compare the impact of carotid artery revascularization on long-term post-operative baroreceptor function and on cognitive brain function, and analyze their influence on clinical outcome. The specific goal is to assess the potential correlation between post-operative autonomic and cognitive function.

2) To assess the solicitation on the carotid wall due to CAS as compared to CEA through structural analysis and mechanical modeling. The specific goal is to assess the potential correlation between stenting, wall damage, baroceptor impairment, and late neurological sequelae. 3) To assess the post-operative carotid hemodynamics combining medical image analysis, clinical data, and computer simulations. The specific goal aims at correlating both local (e.g., wall shear stress (WSS), oscillatory shear index (OSI), relative residence time (RRT)) and global phenomena (controlateral flow, arterial stiffening) with baroreflex function and post-operative neurological outcomes.

Cognitive Assessment. HALO will use existing cognitive assessment infrastructure. Cognitive assessments in our study must take place prior to revascularization or within two weeks after assignment to medical therapy alone. Testing is repeated at 44 days, and every year thereafter up to 4 years. At each test interval, a composite (mean) Z-score is derived from published normative samples for each test outcome. The primary outcome will be at 1 year in which the change in the composite Z-score from baseline will be calculated. Covariates will include age, education and depression. The test battery will be administered the same way for all enrolled patients. The cognitive domains being assessed in HALO are entirely consistent with those encompassed within the NINDS Common Data Elements (CDE).

Imaging protocol. Multimodal MRI, including routine parenchymal sequences and PWI utilizing dynamic susceptibility contrast technique, will be acquired at each participating HALO site. Imaging will take place within 14 days after HALO enrollment and prior to any intervention (carotid artery revascularization).

Standardized contrast agent injection protocol, appropriate preparation, and IV setup is used to ensure good scan quality. An antecubital vein IV catheter of 18-20 gauge is required. A test injection will be performed with approximately 10 ml of normal saline solution.

MRI image acquisition DWI/ADC (b=0, 1000 s/mm2 applied in each of three principal gradient directions), FLAIR, high-resolution T1, and GRE sequences will be acquired on 1.5-3.0 T scanners equipped with echo-planar imaging capability, using standard clinical protocols at participating HALO sites. Total scanning time will be approximately 40 minutes. PWI acquisition protocol will be standardized across all HALO sites, using sequential T2*-weighted (gradient echo) EPI time sequence scanning. A modified 2-phase contrast injection scheme will be used to perform CEMRA and DSC perfusion imaging, without need for additional contrast.

MRI structural analysis. silent infarct --- non-confluent hyperintense lesion >1mm on FLAIR sequence on 1-year MRI not present on baseline FLAIR MRI.

Cerebral microbleed - hypointense 1-2mm non-confluent lesion on baseline GRE sequence.

WMH volume -- White matter hyperintensity volume refers to confluent periventricular high intensity lesions on FLAIR imaging, and will be derived using an automated T2 WMH quantification at the Huston lab.

. Analysis. Specific Aim 1. To determine whether cognition can be improved by revascularization among a subset of HALO patients with hemodynamic changes at baseline.

The primary hypothesis is to assess if the magnitude of the treatment differences (revascularization versus medical management alone) differs between those with flow failure compared to those without flow failure using the Z-scored cognitive outcomes (C0, C(1). That is, the primary hypothesis is an interaction hypothesis that will be assessed using linear regression, specifically: (C1 - C0) = β0 + β1T + β2F + β3TF + β4C0 + (other covariates), where C1 is the cognitive z-score at year 1, C0 the cognitive z-score at baseline, T the treatment indicator variable, F the flow failure indicator variable, and βi the regression parameters to be estimated. The parameter of interest for the primary hypothesis is then β3 that would assess if the magnitude of treatment difference in the change in cognitive score between baseline and 1-year is similar for those with versus without flow failure.

Secondary Aims: To determine if the number of silent infarcts and white matter hyperintensity volume at 1 year is different between the revascularization and the medical-only arms.

For the secondary aims we will calculate the number of new silent cerebral infarctions occurring over the first year, and the change in the WMH volume. The approach for analysis of the number of new silent infarcts will depend on the average number and distribution of the number of new infarcts. The analytic approach will be linear regression if the number of new infarcts is large (considered more likely the case), or Poisson Regression if the number is smaller (considered less likely the case). The analysis of the change in WMH will use a linear regression approach.

ELIGIBILITY:
Inclusion Criteria:

Informed consent signed Patients with >=70% symptomatic or >=80% asymptomatic internal carotid stenosis

Exclusion Criteria:

Incapability to give informed consent Previous disabling stroke Contralateral carotid occlusion or >70% stenosis Systemic disease judged non compatible with the procedures or randomization Suspected or manifested pregnancy General contraindications to MRI or CT studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive score | 1 year
  Among those with flow failure (PWI "time to peak" (TTP) delay>2 sec) and cognitive impairment (>1.0 SD below age-matched norms) at baseline, cognitive change at 1 year will be compared between those receiving revascularization (CEA or CAS) versus those receiving IMM alone.
Change in carotid stenosis | 1 year
  The stenosis of the carotid artery measured by contrast-enhanced CT will be compared between those receiving revascularization (CEA or CAS) versus those receiving IMM alone.
Change in wall shear stress（WSS） | 1 year
  The hemodynamics factors: wall shear stress (WSS) at 1 year will be compared between those receiving revascularization (CEA or CAS) versus those receiving IMM alone.
Change in oscillatory shear index （OSI） | 1 year
  The hemodynamics factors: oscillatory shear index (OSI) at 1 year will be compared between those receiving revascularization (CEA or CAS) versus those receiving IMM alone.
Change in relative residence time（RRT） | 1 year
  The hemodynamics factors: relative residence time (RRT)) at 1 year will be compared between those receiving revascularization (CEA or CAS) versus those receiving IMM alone.

SECONDARY OUTCOMES:
Silent infarcts | 1 year
  MRI-determined silent infarcts present at 1 year that were not present at baseline, comparing by treatment group
White matter hyperintensity (WMH) volume | 1 year
  change in confluent white matter hyperintensity volume at 1 year, comparing by treatment group
Major adverse cardiovascular events | 1 year
  The major adverse cardiovascular events at 1 year, comparing by treatment group
The mortality rate | 1 year
  The mortality rate at 1 year, comparing by treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Cutlip DE, Pinto DS. Extracranial carotid disease revascularization. Circulation. 2012 Nov 27;126(22):2636-44. doi: 10.1161/CIRCULATIONAHA.112.110411. No abstract available. PMID 23184283
- [Background] Auricchio F, Conti M, De Beule M, De Santis G, Verhegghe B. Carotid artery stenting simulation: from patient-specific images to finite element analysis. Med Eng Phys. 2011 Apr;33(3):281-9. doi: 10.1016/j.medengphy.2010.10.011. Epub 2010 Nov 9. PMID 21067964
- [Background] Conti M, Van Loo D, Auricchio F, De Beule M, De Santis G, Verhegghe B, Pirrelli S, Odero A. Impact of carotid stent cell design on vessel scaffolding: a case study comparing experimental investigation and numerical simulations. J Endovasc Ther. 2011 Jun;18(3):397-406. doi: 10.1583/10-3338.1. PMID 21679082
- [Background] Auricchio F, Conti M, Ferrara A, Morganti S, Reali A. Patient-specific finite element analysis of carotid artery stenting: a focus on vessel modeling. Int J Numer Method Biomed Eng. 2013 Jun;29(6):645-64. doi: 10.1002/cnm.2511. Epub 2012 Sep 29. PMID 23729192
- [Background] De Santis G, Conti M, Trachet B, De Schryver T, De Beule M, Degroote J, Vierendeels J, Auricchio F, Segers P, Verdonck P, Verhegghe B. Haemodynamic impact of stent-vessel (mal)apposition following carotid artery stenting: mind the gaps! Comput Methods Biomech Biomed Engin. 2013;16(6):648-59. doi: 10.1080/10255842.2011.629997. Epub 2011 Dec 8. PMID 22149183
- [Background] De Santis G, Trachet B, Conti M, De Beule M, Morbiducci U, Mortier P, Segers P, Verdonck P, Verhegghe B. A computational study of the hemodynamic impact of open- versus closed-cell stent design in carotid artery stenting. Artif Organs. 2013 Jul;37(7):E96-106. doi: 10.1111/aor.12046. Epub 2013 Apr 12. PMID 23578331
- [Background] Hathcock JJ. Flow effects on coagulation and thrombosis. Arterioscler Thromb Vasc Biol. 2006 Aug;26(8):1729-37. doi: 10.1161/01.ATV.0000229658.76797.30. Epub 2006 Jun 1. PMID 16741150
- [Background] Davies PF. Overview: temporal and spatial relationships in shear stress-mediated endothelial signalling. J Vasc Res. 1997 May-Jun;34(3):208-11. doi: 10.1159/000159224. No abstract available. PMID 9226302
- [Background] Bohm M, Cotton D, Foster L, Custodis F, Laufs U, Sacco R, Bath PM, Yusuf S, Diener HC. Impact of resting heart rate on mortality, disability and cognitive decline in patients after ischaemic stroke. Eur Heart J. 2012 Nov;33(22):2804-12. doi: 10.1093/eurheartj/ehs250. Epub 2012 Aug 26. PMID 22922507
- [Background] Irvine CD, Gardner FV, Davies AH, Lamont PM. Cognitive testing in patients undergoing carotid endarterectomy. Eur J Vasc Endovasc Surg. 1998 Mar;15(3):195-204. doi: 10.1016/s1078-5884(98)80176-7. PMID 9587331
- [Background] Hayase H, Tokunaga K, Nakayama T, Sugiu K, Nishida A, Arimitsu S, Hishikawa T, Ono S, Ohta M, Date I. Computational fluid dynamics of carotid arteries after carotid endarterectomy or carotid artery stenting based on postoperative patient-specific computed tomography angiography and ultrasound flow data. Neurosurgery. 2011 Apr;68(4):1096-101; discussion 1101. doi: 10.1227/NEU.0b013e318208f1a0. PMID 21221041
- [Background] Marshall RS, Lazar RM, Liebeskind DS, Connolly ES, Howard G, Lal BK, Huston J 3rd, Meschia JF, Brott TG. Carotid revascularization and medical management for asymptomatic carotid stenosis - Hemodynamics (CREST-H): Study design and rationale. Int J Stroke. 2018 Dec;13(9):985-991. doi: 10.1177/1747493018790088. Epub 2018 Aug 22. PMID 30132751
- [Background] Howard VJ, Meschia JF, Lal BK, Turan TN, Roubin GS, Brown RD Jr, Voeks JH, Barrett KM, Demaerschalk BM, Huston J 3rd, Lazar RM, Moore WS, Wadley VG, Chaturvedi S, Moy CS, Chimowitz M, Howard G, Brott TG; CREST-2 study investigators. Carotid revascularization and medical management for asymptomatic carotid stenosis: Protocol of the CREST-2 clinical trials. Int J Stroke. 2017 Oct;12(7):770-778. doi: 10.1177/1747493017706238. Epub 2017 May 2. PMID 28462683
- [Background] Schroder J, Heinze M, Gunther M, Cheng B, Nickel A, Schroder T, Fischer F, Kessner SS, Magnus T, Fiehler J, Larena-Avellaneda A, Gerloff C, Thomalla G. Dynamics of brain perfusion and cognitive performance in revascularization of carotid artery stenosis. Neuroimage Clin. 2019;22:101779. doi: 10.1016/j.nicl.2019.101779. Epub 2019 Mar 13. PMID 30903966
- [Background] Piegza M, Wieckiewicz G, Wierzba D, Piegza J. Cognitive Functions in Patients after Carotid Artery Revascularization-A Narrative Review. Brain Sci. 2021 Oct 1;11(10):1307. doi: 10.3390/brainsci11101307. PMID 34679372